CLINICAL TRIAL: NCT01438983
Title: Evaluation the Effect of Dietary Type on Oral Candida Carriage in Infants
Brief Title: Oral Candida in Infants and Dietary Type
Status: Completed | Type: Observational
Sponsor: Shahid Sadoughi University of Medical Sciences and Health Services (Other)
Responsible Party: Principal Investigator, Nastaran Azimi, Principal Investigator, Shahid Sadoughi University of Medical Sciences and Health Services
Other Study IDs: uni43
Record Dates: First submitted 2011-09-18; First posted 2011-09-22 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Oral Candida; Breastfeeding; Bottle Feeding
MeSH Terms: conditions — Candidiasis; Breast Feeding; Bottle Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — infants with unremarkable health histories, normal weight, free of sign or symptom of oral candidiasis or other mucosal disease.their mothers were also healthy and without sign or symptom of vagina or mammary candidiasis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- breastfeeding infants
- bottle feeding infants

SUMMARY:
This is an observational, non-randomised trial to evaluate the effect of dietary type on infants oral candida colonization the investigators evaluated 90 infants in 1-24 months (45 breastfeeding and 45 bottle feeding infants) who attended to Yazd clinic for regular pediatric appointment. Infants with unremarkable health histories, normal weight, free of sign or symptom of oral candidiasis or other mucosal disease. Their mothers were also healthy and without sign or symptom of vagina or mammary candidiasis. Pacifier usage, use of antibiotics in last months, sign or symptom of oral candidiasis in infants or vagina and mammary candidiasis in mothers were exclusion criteria.

DETAILED DESCRIPTION:
After filling in a questionnaire about infants dietary intake, age and sex and their mothers education level and health condition, a pre-moistened sterile cotton swab was taken from dorsal surface of tongue and mid-plate. The swabs were cultured in agar plate containing sabourauds dextrose agar medium with chloramphenicol, and kept in 37 C for 48 hours. The number of candida colonies was counted and germ tube test performed to separate candida albicans from other types. The data was collected and analyzed by SPSS software and chi-square, logistic regression and mann-whitney test. Study hypothesis: feeding by mothers milk reduces oral candida colonization.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants
* healthy mothers

Exclusion Criteria:

* pacifier usage
* use of antibiotics in last month
* sign or symptom of oral candidiasis in infants
* vagina and mammary candidiasis in mothers

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators evaluated 90 infants in 1-24 months (45 breastfeeding and 45 bottle feeding infants) who attended to Yazd nikoopur clinic for regular pediatric appointment.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-07; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
mean number of candida colonies | 6 months
  number of candida colonies growth in agar plate

SECONDARY OUTCOMES:
prevalence of oral candida colonization in infants according to age and sex | 6 months
  exist of candida colony in agar plate

CONTACTS AND LOCATIONS:
Overall Officials: nastaran azimi, dr, Principal Investigator — shahid sadoughi university of medical sciences and health science
Locations (1):
- Nastaran Azimi, Yazd, Yazd Province, Iran